CLINICAL TRIAL: NCT04564339
Title: A Phase 2, Double-Blind, Randomized, Placebo-Controlled Study to Evaluate the Efficacy and Safety of Ravulizumab in Adult Participants With Proliferative Lupus Nephritis (LN) or Immunoglobulin A Nephropathy (IgAN)
Brief Title: Study of Ravulizumab in Proliferative Lupus Nephritis (LN) or Immunoglobulin A Nephropathy (IgAN)
Acronym: SANCTUARY
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor Decision.
Sponsor: Alexion Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ALXN1210-NEPH-202; 2020-001537-13 (EudraCT Number)
Record Dates: First submitted 2020-09-21; First posted 2020-09-25 (Actual); Results first posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Lupus Nephritis; Immunoglobulin A Nephropathy
Keywords: glomerulonephritis; IGA; lupus nephritis; complement C5
MeSH Terms: conditions — Lupus Nephritis; Glomerulonephritis, IGA; Glomerulonephritis | interventions — ravulizumab

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Participants, all investigative site personnel, and any Alexion employee, or designee, directly associated with the conduct of the study will be blinded to participant treatment assignments during the 26-week Initial Evaluation Period. Both the participants and the investigative site personnel will remain blinded for the remaining 24-week Extension Period.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Ravulizumab: LN Cohort (Experimental): Eligible participants will receive ravulizumab IV infusion in combination with background therapy during both the Initial Evaluation Period (26 weeks) and Extension Period (24 weeks). During the Follow-up Period (36 weeks) participants will receive background therapy according to the standard of care.
  Interventions: Drug: Ravulizumab; Other: Background Therapy
- Placebo: LN Cohort (Placebo Comparator): Eligible participants will receive placebo IV infusion in combination with background therapy during both the Initial Evaluation Period (26 weeks) and Extension Period (24 weeks). During the Follow-up Period (36 weeks) participants will receive background therapy according to the standard of care.
  Interventions: Drug: Placebo; Other: Background Therapy
- Ravulizumab: IgAN Cohort (Experimental): Eligible participants will receive ravulizumab IV infusion in combination with background therapy during both the Initial Evaluation Period (26 weeks) and Extension Period (24 weeks). During the Follow-up Period (36 weeks) participants will receive background therapy according to the standard of care.
  Interventions: Drug: Ravulizumab; Other: Background Therapy
- Placebo: IgAN Cohort (Placebo Comparator): Eligible participants will receive placebo IV infusion in combination with background therapy during the Initial Evaluation Period (26 weeks) and will switch to ravulizumab for the Extension Period (24 weeks). During the Follow-up Period (36 weeks) participants will receive background therapy according to the standard of care.
  Interventions: Drug: Ravulizumab; Drug: Placebo; Other: Background Therapy

INTERVENTIONS:
Drug: Ravulizumab — Dosages (loading and maintenance) will be based on the participant's body weight.
  Other Names: Ultomiris
  Arms: Placebo: IgAN Cohort; Ravulizumab: IgAN Cohort; Ravulizumab: LN Cohort
Drug: Placebo — Dosages (loading and maintenance) will be based on the participant's body weight.
  Arms: Placebo: IgAN Cohort; Placebo: LN Cohort
Other: Background Therapy — Participants will receive background therapy consistent with the standard of care.

SUMMARY:
The objectives of this study are to evaluate the safety and efficacy of ravulizumab administered by intravenous (IV) infusion compared to placebo and demonstrate proof-of-concept of the efficacy of terminal complement inhibition in participants with LN (LN Cohort) or IgAN (IgAN Cohort).

DETAILED DESCRIPTION:
This study consists of a 6-week Screening Period, 26-week Initial Evaluation Period, a 24-week Extension Period, and a 36-week post-treatment Follow-up Period.

ELIGIBILITY:
Inclusion Criteria:

Common to both disease cohorts:

* Proteinuria ≥1 (gram [g]/day or g/g)
* Vaccinated against meningococcal infection
* Vaccinated for Haemophilus influenzae type b (Hib) and Streptococcus pneumoniae according to national/local regulatory requirements

For LN cohort:

* Diagnosis of active focal or diffuse proliferative LN Class III or IV
* Clinically active LN, requiring/receiving immunosuppression induction treatment

For IgAN cohort:

* Diagnosis of primary IgAN
* Compliance with stable and optimal dose of renin-angiotensin system inhibitor treatment for ≥ 3 months

Exclusion Criteria:

Common to both disease cohorts:

* eGFR < 30 milliliters/minute/1.73 meters squared
* Previously received a complement inhibitor (for example, eculizumab)
* Concomitant significant renal disease other than LN or IgAN
* History of other solid organ or bone marrow transplant
* Uncontrolled hypertension

For IgAN cohort:

* Diagnosis of rapid progressive glomerulonephritis
* Prednisone or prednisone equivalent > 20 milligram (mg) per day for > 14 consecutive days or any other immunosuppression within 6 months

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 123 (Actual)
Dates: Start 2021-01-19 (Actual); Primary Completion 2025-03-26 (Actual); Study Completion 2025-08-18 (Actual)

CONTACTS AND LOCATIONS:
Locations (55):
- United States (16):
  - Research Site, San Dimas, California
  - Research Site, Santa Monica, California
  - Research Site, South Gate, California
  - Research Site, Stanford, California
  - Research Site, Orlando, Florida
  - Research Site, Plantation, Florida
  - Research Site, Lawrenceville, Georgia
  - Research Site, Lexington, Kentucky
  - Research Site, Louisville, Kentucky
  - Research Site, Boston, Massachusetts
  - Research Site, Kansas City, Missouri
  - Research Site, New York, New York
  - Research Site, Chapel Hill, North Carolina
  - Research Site, Columbus, Ohio
  - Research Site, El Paso, Texas
  - Research Site, Houston, Texas
- Australia (3):
  - Research Site, Herston
  - Research Site, Parkville
  - Research Site, Westmead
- Canada (3):
  - Research Site, London, Ontario
  - Research Site, Montreal, Quebec
  - Research Site, Québec, Quebec
- France (6):
  - Research Site, Clermont-Ferrand
  - Research Site, Le Kremlin-Bicêtre
  - Research Site, Paris
  - Research Site, Saint-Priest-en-Jarez
  - Research Site, Strasbourg
  - Research Site, Toulouse
- Germany (4):
  - Research Site, Berlin
  - Research Site, Essen
  - Research Site, Hanover
  - Research Site, Lübeck
- Italy (4):
  - Research Site, Bologna
  - Research Site, Brescia
  - Research Site, Florence
  - Research Site, Torino
- Research Site, Maastricht, Netherlands
- Research Site, Lodz, Poland
- South Korea (3):
  - Research Site, Anyang-si
  - Research Site, Seongnam-si
  - Research Site, Seoul
- Spain (8):
  - Research Site, Barcelona
  - Research Site, Lleida
  - Research Site, Madrid
  - Research Site, Málaga
  - Research Site, Palma de Mallorca
  - Research Site, Seville
  - Research Site, Valencia
  - Research Site, Zaragoza
- Taiwan (3):
  - Research Site, Kaohsiung City
  - Research Site, New Taipei City
  - Research Site, Taichung
- United Kingdom (3):
  - Research Site, Edgbaston
  - Research Site, London
  - Research Site, Salford

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lafayette R, Tumlin J, Fenoglio R, Kaufeld J, Perez Valdivia MA, Wu MS, Susan Huang SH, Alamartine E, Kim SG, Yee M, Kateifides A, Rice K, Garlo K, Barratt J; SANCTUARY Study Investigators. Efficacy and Safety of Ravulizumab in IgA Nephropathy: A Phase 2 Randomized Double-Blind Placebo-Controlled Trial. J Am Soc Nephrol. 2025 Apr 1;36(4):645-656. doi: 10.1681/ASN.0000000534. Epub 2024 Oct 25. PMID 39455063
- [Derived] Avasare R, Drexler Y, Caster DJ, Mitrofanova A, Jefferson JA. Management of Lupus Nephritis: New Treatments and Updated Guidelines. Kidney360. 2023 Oct 1;4(10):1503-1511. doi: 10.34067/KID.0000000000000230. PMID 37528520
- See also: Related Info — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=ALXN1210-NEPH-202&attachmentIdentifier=9837083f-ecf8-4776-a44c-5c0c5df940f9&fileName=ALXN1210-NEPH-202_IgAN_Cohort_Final_Analysis_Combined_2_CSR_Synopsis_(Final)_Redacted.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: For the lupus nephritis (LN) cohort, a total of 57 participants were enrolled in the study and randomized. For the immunoglobulin A nephropathy (IgAN) cohort, a total of 66 participants were enrolled in the study and randomized.
Groups:
- LN Cohort: Ravulizumab: Participants with LN received body weight-based loading dose of ravulizumab intravenous (IV) infusion on Day 1, followed by body weight-based maintenance doses of ravulizumab on Day 15 and then every 8 weeks (q8w) thereafter during the Initial Evaluation Period (26 weeks). Participants continued on the same maintenance regimen during the Extension Period (24 weeks).
- LN Cohort: Placebo: Participants with LN received a loading dose of ravulizumab matched placebo IV infusion on Day 1, followed by maintenance doses of ravulizumab matched placebo on Day 15 and then q8w thereafter during both the Initial Evaluation Period (26 weeks). Participants continued on the same maintenance doses of ravulizumab matched placebo during the Extension Period (24 weeks).
- IgAN Cohort: Ravulizumab: Participants with IgAN received body weight-based loading dose of ravulizumab IV infusion on Day 1, followed by body weight-based maintenance doses of ravulizumab on Day 15 and then q8w thereafter during both the Initial Evaluation Period (26 weeks). Participants received a blinded dose of ravulizumab at Week 26 and then open-label body weight-based dosing of ravulizumab q8w until the end of the Extension Period (24 weeks).
- IgAN Cohort: Placebo: Participants with IgAN received a loading dose of ravulizumab matched placebo IV infusion on Day 1, followed by maintenance doses of ravulizumab matched placebo on Day 15 and then q8w thereafter during both the Initial Evaluation Period (26 weeks). Participants switched to receive a blinded loading dose of ravulizumab at Week 26 and then open-label body weight-based dosing of ravulizumab q8w until the end of the Extension Period (24 weeks).
Period: Initial Evaluation Period (26 Weeks)
Arm/Group | LN Cohort: Ravulizumab | LN Cohort: Placebo | IgAN Cohort: Ravulizumab | IgAN Cohort: Placebo
Started | 38 | 19 | 43 | 23
Received at Least 1 Dose of Study Drug | 38 | 19 | 43 | 23
Completed | 36 | 18 | 42 | 23
Not Completed | 2 | 1 | 1 | 0
Not completed — Withdrawal by Subject | 1 | 1 | 1 | 0
Not completed — Physician Decision | 1 | 0 | 0 | 0
Period: Extension Period (Week 26 to Week 50)
Arm/Group | LN Cohort: Ravulizumab | LN Cohort: Placebo | IgAN Cohort: Ravulizumab | IgAN Cohort: Placebo
Started | 36 | 18 | 42 | 23
Completed | 34 | 17 | 41 | 23
Not Completed | 2 | 1 | 1 | 0
Not completed — Physician Decision | 1 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0
Not completed — Study Terminated by Sponsor | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS) included all randomized participants who received at least 1 dose of the study intervention.
Groups:
- LN Cohort: Ravulizumab: Participants with LN received body weight-based loading dose of ravulizumab IV infusion on Day 1, followed by body weight-based maintenance doses of ravulizumab on Day 15 and then q8w thereafter during the Initial Evaluation Period (26 weeks). Participants continued on the same maintenance regimen during the Extension Period (24 weeks).
- Total: Total of all reporting groups
Arm/Group | LN Cohort: Ravulizumab | LN Cohort: Placebo | IgAN Cohort: Ravulizumab | IgAN Cohort: Placebo | Total
Number analyzed (Participants) | 38 | 19 | 43 | 23 | 123
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 38 | 18 | 43 | 22 | 121
  >=65 years | 0 | 1 | 0 | 1 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 15 | 22 | 8 | 72
  Male | 11 | 4 | 21 | 15 | 51
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 5 | 11 | 3 | 22
  Not Hispanic or Latino | 31 | 14 | 27 | 20 | 92
  Unknown or Not Reported | 4 | 0 | 5 | 0 | 9
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Asian | 13 | 8 | 7 | 7 | 35
  Race: Black or African American | 6 | 1 | 0 | 0 | 7
  Race: Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 0 | 1
  Race: White | 14 | 5 | 31 | 16 | 66
  Race: Asian, White | 1 | 0 | 0 | 0 | 1
  Race: Not Reported | 3 | 1 | 4 | 0 | 8
  Race: Unknown | 1 | 2 | 0 | 0 | 3
  Race: Other | 0 | 1 | 1 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: IgAN Cohort: Percentage Change From Baseline in Proteinuria at Week 26 Measured by Absolute Protein (Based on 24-hour Urine Collections)
Description: Proteinuria, the presence of excess proteins in the urine, was measured by absolute protein in grams/day derived from 24-hour urine collections obtained at designated timepoints. A negative change from baseline indicated a reduction in symptoms.
Time Frame: Baseline, Week 26
Population: FAS included all randomized participants who received at least 1 dose of the study intervention. 'Overall number of participants analyzed' = participants evaluable for this outcome measure.
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: percentage change
Arm/Group | IgAN Cohort: Ravulizumab | IgAN Cohort: Placebo
Number analyzed (Participants) | 41 | 22
percentage change | -41.9 [-50.2 to -32.0] | -16.8 [-31.8 to 1.6]
Statistical Analysis 1: Comparison: IgAN Cohort: Ravulizumab vs IgAN Cohort: Placebo; Test type: Superiority; p = 0.0053, ANCOVA; Percentage Difference = -30.1, 90% CI 2-sided [-43.5 to -13.7]

2. Primary Outcome: LN Cohort: Percentage Change From Baseline in Proteinuria at Week 26 Measured by Urine Protein to Creatinine Ratio (UPCR) (Based on 24-hour Urine Collections)
Description: Proteinuria, the presence of excess proteins in the urine, was measured by UPCR in grams/gram derived from 24-hour urine collections obtained at designated timepoints. A negative change from baseline indicated a reduction in symptoms.
Time Frame: Baseline, Week 26
Population: as for outcome 1
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: percentage change
Arm/Group | LN Cohort: Ravulizumab | LN Cohort: Placebo
Number analyzed (Participants) | 33 | 18
percentage change | -69.7 [-79.9 to -54.5] | -67.0 [-80.8 to -43.1]
Statistical Analysis 1: Comparison: LN Cohort: Ravulizumab vs LN Cohort: Placebo; Test type: Superiority; p = 0.8036, ANCOVA; Percentage Difference = -8.4, 90% CI 2-sided [-48.6 to 63.2]

3. Secondary Outcome: IgAN Cohort: Percentage Change From Baseline in Proteinuria at Week 50 Measured by Absolute Protein (Based on 24-hour Urine Collections)
Description: as for outcome 1
Time Frame: Baseline, Week 50
Population: as for outcome 1
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: percentage change
Groups:
- IgAN Cohort - Ravulizumab: Participants with immunoglobulin A nephropathy (IgAN) received a body weight-based loading dose of ravulizumab IV infusion on Day 1, followed by body weight-based maintenance doses of ravulizumab on Day 15 and then q8w thereafter during both the Initial Evaluation Period (26 weeks). Participants received a blinded dose of ravulizumab at Week 26 and then open-label body weight-based dosing of ravulizumab q8w until the end of the Extension Period (24 weeks).
- IgAN Cohort - Placebo: Participants with IgAN received a loading dose of ravulizumab matched placebo IV infusion on Day 1, followed by maintenance doses of ravulizumab matched placebo on Day 15 and then q8w thereafter during both the Initial Evaluation Period (26 weeks). Participants switched to receive a blinded loading dose of ravulizumab at Week 26 and then open-label body weight-based dosing of ravulizumab q8w until the end of the Extension Period (24 weeks).
Arm/Group | IgAN Cohort - Ravulizumab | IgAN Cohort - Placebo
Number analyzed (Participants) | 41 | 23
percentage change | -44.8 [-55.1 to -32.1] | -45.1 [-58.0 to -28.4]

4. Secondary Outcome: LN Cohort: Percentage Change From Baseline in Proteinuria at Week 50 Measured by UPCR (Based on 24-hour Urine Collections)
Description: as for outcome 2
Time Frame: Baseline, Week 50
Population: as for outcome 1
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: percentage change
Arm/Group | LN Cohort: Ravulizumab | LN Cohort: Placebo
Number analyzed (Participants) | 30 | 14
percentage change | -77.1 [-86.0 to -62.4] | -75.0 [-87.2 to -51.2]

5. Secondary Outcome: IgAN Cohort: Percentage of Participants With > 30% and > 50% Reduction in Proteinuria at Week 26 and Week 50 Compared to Baseline Assessed Using 24-hour Urine Collections
Description: Proteinuria, the presence of excess proteins in the urine, was measured by absolute protein in grams/day derived from 24-hour urine collections obtained at designated timepoints.
Time Frame: Baseline to Week 26 and Week 50
Population: FAS included all randomized participants who received at least 1 dose of the study intervention. 'Overall number of participants analyzed' = participants evaluable for this outcome measure. 'Number analyzed' = participants evaluable at specified timepoint.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | IgAN Cohort: Ravulizumab | IgAN Cohort: Placebo
Number analyzed (Participants) | 41 | 23
percentage of participants
  Week 26: >30% Reduction: number analyzed (Participants) | 41 | 22
  Week 26: >30% Reduction | 68.3 [51.9 to 81.9] | 40.9 [20.7 to 63.6]
  Week 26: >50% Reduction: number analyzed (Participants) | 41 | 22
  Week 26: >50% Reduction | 43.9 [28.5 to 60.3] | 18.2 [5.2 to 40.3]
  Week 50: >30% Reduction | 63.4 [46.9 to 77.9] | 60.9 [38.5 to 80.3]
  Week 50: >50% Reduction | 36.6 [22.1 to 53.1] | 39.1 [19.7 to 61.5]

6. Secondary Outcome: LN Cohort: Percentage of Participants With > 30% and > 50% Reduction in Proteinuria at Week 26 and Week 50 Compared to Baseline Assessed Using 24-hour Urine Collections
Description: Proteinuria, the presence of excess proteins in the urine, was measured by UPCR in grams/gram derived from 24-hour urine collections obtained at designated timepoints.
Time Frame: Baseline to Week 26 and Week 50
Population: FAS included all randomized participants who received at least 1 dose of the study intervention.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | LN Cohort: Ravulizumab | LN Cohort: Placebo
Number analyzed (Participants) | 38 | 19
percentage of participants
  Week 26: >30% Reduction | 50.0 [33.4 to 66.6] | 73.7 [48.8 to 90.9]
  Week 26: >50% Reduction | 47.4 [31.0 to 64.2] | 57.9 [33.5 to 79.7]
  Week 50: >30% Reduction | 55.3 [38.3 to 71.4] | 63.2 [38.4 to 83.7]
  Week 50: >50% Reduction | 52.6 [35.8 to 69.0] | 47.4 [24.4 to 71.1]

7. Secondary Outcome: IgAN Cohort: Change From Baseline in Estimated Glomerular Filtration Rate (eGFR) at Week 26 and Week 50
Description: Changes in kidney function were monitored using measurements of eGFR and calculated based on the Chronic Kidney Disease Epidemiology Collaboration formula. Results are reported in milliliters/minute/1.73 meters squared (mL/min/1.73 m^2). Estimates of change from baseline are least-square means based on a mixed-effect model for repeated measures model that included change from baseline as the response variable, treatment as independent variable and adjusts for covariates of baseline and the stratification factor at randomization. An increase in eGFR in response to treatment indicated a reduction in symptoms.
Time Frame: Baseline, Week 26 and Week 50
Population: as for outcome 5
Measure: Least Squares Mean (95% Confidence Interval); unit: mL/min/1.73 m^2
Arm/Group | IgAN Cohort: Ravulizumab | IgAN Cohort: Placebo
Number analyzed (Participants) | 42 | 23
mL/min/1.73 m^2
  Change at Week 26 | 0.22 [-2.30 to 2.74] | -4.51 [-7.90 to -1.11]
  Change at Week 50: number analyzed (Participants) | 41 | 23
  Change at Week 50 | -3.87 [-6.41 to -1.33] | -6.33 [-9.72 to -2.94]

8. Secondary Outcome: LN Cohort: Change From Baseline in eGFR at Week 26 and Week 50
Description: Changes in kidney function were monitored using measurements of eGFR and calculated based on the Chronic Kidney Disease Epidemiology Collaboration formula. Results are reported in mL/min/1.73 m^2. Estimates of change from baseline are least-square means based on a mixed-effect model for repeated measures model that included change from baseline as the response variable, treatment as independent variable and adjusts for covariates of baseline and the stratification factor at randomization. An increase in eGFR in response to treatment indicated a reduction in symptoms.
Time Frame: Baseline, Week 26 and Week 50
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mL/min/1.73 m^2
Arm/Group | LN Cohort: Ravulizumab | LN Cohort: Placebo
Number analyzed (Participants) | 32 | 17
mL/min/1.73 m^2
  Change at Week 26 | 11.59 (3.38) | 14.04 (4.56)
  Change at Week 50: number analyzed (Participants) | 30 | 15
  Change at Week 50 | 12.12 (3.49) | 14.83 (4.86)

9. Secondary Outcome: IgAN Cohort: Change From Baseline in Serum Complement Component 3 (C3) and Complement Component 4 (C4) Concentrations at Week 26 and Week 50
Time Frame: Baseline, Week 26 and Week 50
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: grams/liter
Arm/Group | IgAN Cohort: Ravulizumab | IgAN Cohort: Placebo
Number analyzed (Participants) | 42 | 22
grams/liter
  C3: Change at Week 26 | 0.027 (0.2389) | -0.019 (0.2366)
  C3: Change at Week 50: number analyzed (Participants) | 41 | 20
  C3: Change at Week 50 | -0.001 (0.1902) | -0.084 (0.1861)
  C4: Change at Week 26 | -0.005 (0.0576) | -0.001 (0.0566)
  C4: Change at Week 50: number analyzed (Participants) | 41 | 20
  C4: Change at Week 50 | -0.006 (0.0510) | -0.027 (0.0489)

10. Secondary Outcome: LN Cohort: Change From Baseline in Serum C3 and C4 Concentrations at Week 26 and Week 50
Time Frame: Baseline, Week 26 and Week 50
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: grams/liter
Arm/Group | LN Cohort: Ravulizumab | LN Cohort: Placebo
Number analyzed (Participants) | 36 | 17
grams/liter
  C3: Change at Week 26 | 0.139 (0.2414) | 0.130 (0.1809)
  C3: Change at Week 50: number analyzed (Participants) | 34 | 17
  C3: Change at Week 50 | 0.213 (0.4783) | 0.247 (0.2703)
  C4: Change at Week 26 | 0.041 (0.0775) | 0.028 (0.0668)
  C4: Change at Week 50: number analyzed (Participants) | 34 | 17
  C4: Change at Week 50 | 0.042 (0.0887) | 0.052 (0.0891)

11. Secondary Outcome: LN Cohort: Percentage of Participants Meeting the Criteria for Complete Renal Response (CRR)
Description: The CRR was defined as meeting all 3 of the following criteria: - UPCR ≤0.5 gram/gram (g/g); - eGFR >60 mL/min/1.73 m^2 or no eGFR reduction ≥20% from baseline; and - no treatment failure. Treatment failure was defined as the receipt of additional standard of care therapy at any time during the study for protocol-defined renal flare, severe extrarenal systemic lupus erythematosus (SLE) flare, or suboptimal response.
Time Frame: Week 26 and Week 50
Population: FAS included all randomized participants who received at least 1 dose of the study intervention.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | LN Cohort: Ravulizumab | LN Cohort: Placebo
Number analyzed (Participants) | 38 | 19
percentage of participants
  Week 26 | 26.3 [13.4 to 43.1] | 21.1 [6.1 to 45.6]
  Week 50 | 42.1 [26.3 to 59.2] | 31.6 [12.6 to 56.6]

12. Secondary Outcome: LN Cohort: Percentage of Participants Meeting the Criteria for Partial Renal Response (PRR)
Description: The PRR was defined as meeting all 3 of the following criteria: - decrease of UPCR >50% from baseline; - eGFR >60 mL/min/1.73 m^2 or no eGFR reduction ≥20% from baseline; and - no treatment failure. Treatment failure was defined as the receipt of additional standard of care therapy at any time during the study for protocol-defined renal flare, severe extrarenal SLE flare, or suboptimal response.
Time Frame: Week 26 and Week 50
Population: FAS included all randomized participants who received at least 1 dose of the study intervention.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | LN Cohort: Ravulizumab | LN Cohort: Placebo
Number analyzed (Participants) | 38 | 19
percentage of participants
  Week 26 | 15.8 [6.0 to 31.3] | 36.8 [16.3 to 61.6]
  Week 50 | 10.5 [2.9 to 24.8] | 10.5 [1.3 to 33.1]

13. Secondary Outcome: LN Cohort: Time to Urine Protein to Creatinine Ratio (UPCR) < 0.5 g/g, as Measured by Spot Urine Samples
Time Frame: Baseline through Week 50
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | LN Cohort: Ravulizumab | LN Cohort: Placebo
Number analyzed (Participants) | 36 | 18
days | 184.0 [71.0 to NA] — Due to insufficient number of participants with response, upper limit of 95% confidence interval (CI) could not be estimated. | 295.0 [128.0 to NA] — Due to insufficient number of participants with response, upper limit of 95% CI could not be estimated.

14. Secondary Outcome: LN Cohort: Percentage of Participants Achieving Corticosteroid Taper to 7.5 Milligrams (mg)/Day
Description: A corticosteroid taper was carried out per protocol at the clinical discretion of the investigator.
Time Frame: Week 14, Week 26, and Week 50
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | LN Cohort: Ravulizumab | LN Cohort: Placebo
Number analyzed (Participants) | 38 | 18
percentage of participants
  Week 14 | 84.2 [68.7 to 94.0] | 94.4 [72.7 to 99.9]
  Week 26: number analyzed (Participants) | 36 | 18
  Week 26 | 94.4 [81.3 to 99.3] | 100 [81.5 to 100]
  Week 50: number analyzed (Participants) | 34 | 17
  Week 50 | 76.5 [58.8 to 89.3] | 82.4 [56.6 to 96.2]

15. Secondary Outcome: LN Cohort: Percentage of Participants With Renal Flare
Description: Renal flare was determined in the opinion of the investigator and additional protocol-specified criteria. For participants who achieved a CRR, a renal flare was the reproducible recurrence of proteinuria ≥1g/g. For all other participants, a renal flare was either of the following: a reproducible increase of serum creatinine >25% higher than baseline, above the upper limit of normal (plus additional protocol-specified criteria), or a reproducible doubling of the UPCR from a 24-hour urine collection compared with the lowest previous value obtained after the first dose of study intervention.
Time Frame: Baseline through Week 50
Population: FAS included all randomized participants who received at least 1 dose of the study intervention.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | LN Cohort: Ravulizumab | LN Cohort: Placebo
Number analyzed (Participants) | 38 | 19
percentage of participants | 13.2 [4.4 to 28.1] | 5.3 [0.1 to 26.0]

16. Secondary Outcome: LN Cohort: Percentage of Participants With Extrarenal Systemic Lupus Erythematosus (SLE) Flare
Description: Extrarenal SLE flare was defined as an increase in the Systemic Lupus Erythematosus Disease Activity Index 2000 (SLEDAI-2K) Safety of Estrogens in Lupus Erythematosus National Assessment modification ≥4 points that was not accounted for by proteinuria, hematuria, urinary cellular casts, hypocomplementemia, or an increase in anti-double-stranded DNA antibody level. The SLEDAI-2K is an instrument that was used to assess the disease activity of extrarenal SLE flare across 18 disease descriptors. Each descriptor carried a weighted value ranging from 1-8, with the reported score calculated as the sum of these descriptors and ranging from 0 to 85. Higher scores represent increased degrees of disease activity.
Time Frame: Baseline through Week 50
Population: FAS included all randomized participants who received at least 1 dose of the study intervention.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | LN Cohort: Ravulizumab | LN Cohort: Placebo
Number analyzed (Participants) | 38 | 19
percentage of participants | 2.6 [0.1 to 13.8] | 0.0 [0.0 to 17.6]

17. Secondary Outcome: LN Cohort: Percentage of Participants With Treatment Failure
Description: Treatment failure was defined as the receipt of additional standard of care therapy at any time during the study for protocol-defined renal flare, severe extrarenal SLE flare, or suboptimal response.
Time Frame: Baseline through Week 50
Population: FAS included all randomized participants who received at least 1 dose of the study intervention.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | LN Cohort: Ravulizumab | LN Cohort: Placebo
Number analyzed (Participants) | 38 | 19
percentage of participants | 26.3 [13.4 to 43.1] | 10.5 [1.3 to 33.1]

18. Secondary Outcome: LN Cohort: Percentage of Participants With Suboptimal Response
Description: A suboptimal response was to be determined in the opinion of the investigator in addition to the following criterion: reproducible proteinuria ≤25% decreased compared to baseline based on UPCR on a 24-hour urine collection performed by a central laboratory.
Time Frame: Baseline through Week 50
Population: FAS included all randomized participants who received at least 1 dose of the study intervention.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | LN Cohort: Ravulizumab | LN Cohort: Placebo
Number analyzed (Participants) | 38 | 19
percentage of participants | 7.9 [1.7 to 21.4] | 10.5 [1.3 to 33.1]

19. Secondary Outcome: LN Cohort: Change From Baseline in Serum Albumin at Week 26 and Week 50
Description: For the determination of serum albumin, blood samples were obtained at designated time points.
Time Frame: Baseline, Week 26, Week 50
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: grams/liter
Arm/Group | LN Cohort: Ravulizumab | LN Cohort: Placebo
Number analyzed (Participants) | 35 | 18
grams/liter
  Change at Week 26 | 5.14 (5.048) | 6.94 (5.252)
  Change at Week 50: number analyzed (Participants) | 34 | 17
  Change at Week 50 | 6.44 (6.761) | 10.65 (5.408)

20. Secondary Outcome: IgAN Cohort: Percentage of Participants Meeting the Criteria for Partial Remission
Description: Partial remission was defined as mean proteinuria <1 g/24 hours, based on two valid 24-hour urine collections obtained within 2 weeks prior to the study visit.
Time Frame: Week 26 and Week 50
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | IgAN Cohort: Ravulizumab | IgAN Cohort: Placebo
Number analyzed (Participants) | 41 | 23
percentage of participants
  Week 26: number analyzed (Participants) | 41 | 22
  Week 26 | 26.8 [14.2 to 42.9] | 18.2 [5.2 to 40.3]
  Week 50 | 39.0 [24.2 to 55.5] | 26.1 [10.2 to 48.4]

ADVERSE EVENTS:
Time Frame: Baseline up to Week 86
Description: Safety Set included all participants who received at least 1 dose of study intervention.
Groups:
- Initial Evaluation Period: LN Cohort - Ravulizumab: Participants with LN received body weight-based loading dose of ravulizumab IV infusion on Day 1, followed by body weight-based maintenance doses of ravulizumab on Day 15 and then q8w thereafter during the Initial Evaluation Period (26 weeks).
- Initial Evaluation Period: LN Cohort - Placebo: Participants with LN received a loading dose of ravulizumab matched placebo IV infusion on Day 1, followed by maintenance doses of ravulizumab matched placebo on Day 15 and then q8w thereafter during both the Initial Evaluation Period (26 weeks).
- Initial Evaluation Period: IgAN Cohort - Ravulizumab: Participants with immunoglobulin A nephropathy (IgAN) received body weight-based loading dose of ravulizumab IV infusion on Day 1, followed by body weight-based maintenance doses of ravulizumab on Day 15 and then q8w thereafter during both the Initial Evaluation Period (26 weeks).
- Initial Evaluation Period: IgAN Cohort - Placebo: Participants with IgAN received a loading dose of ravulizumab matched placebo IV infusion on Day 1, followed by maintenance doses of ravulizumab matched placebo on Day 15 and then q8w thereafter during both the Initial Evaluation Period (26 weeks).
- Extension Period: LN Cohort - Ravulizumab to Ravulizumab: Participants continued on the same maintenance regimen (as received during the Initial Evaluation Period) during the Extension Period (24 weeks).
- Extension Period: LN Cohort - Placebo to Placebo: Participants continued to receive ravulizumab matched placebo q8w until the end of the Extension Period (24 weeks).
- Extension Period: IgAN Cohort - Ravulizumab to Ravulizumab: Participants received a blinded dose of ravulizumab at Week 26 and then open-label body weight-based dosing of ravulizumab q8w until the end of the Extension Period (24 weeks).
- Extension Period: IgAN Cohort - Placebo to Ravulizumab: Participants switched to receive a blinded loading dose of ravulizumab at Week 26 and then open-label body weight-based dosing of ravulizumab q8w until the end of the Extension Period (24 weeks).
Arm/Group | Initial Evaluation Period: LN Cohort - Ravulizumab | Initial Evaluation Period: LN Cohort - Placebo | Initial Evaluation Period: IgAN Cohort - Ravulizumab | Initial Evaluation Period: IgAN Cohort - Placebo | Extension Period: LN Cohort - Ravulizumab to Ravulizumab | Extension Period: LN Cohort - Placebo to Placebo | Extension Period: IgAN Cohort - Ravulizumab to Ravulizumab | Extension Period: IgAN Cohort - Placebo to Ravulizumab
All-Cause Mortality (participants affected / at risk) | 0/38 | 0/19 | 0/43 | 0/23 | 0/36 | 0/18 | 0/42 | 0/23
Serious Adverse Events (participants affected / at risk) | 6/38 | 2/19 | 1/43 | 0/23 | 6/36 | 2/18 | 0/42 | 0/23
Other Adverse Events (participants affected / at risk) | 28/38 | 15/19 | 17/43 | 9/23 | 14/36 | 16/18 | 11/42 | 2/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Initial Evaluation Period: LN Cohort - Ravulizumab (N=38) | Initial Evaluation Period: LN Cohort - Placebo (N=19) | Initial Evaluation Period: IgAN Cohort - Ravulizumab (N=43) | Initial Evaluation Period: IgAN Cohort - Placebo (N=23) | Extension Period: LN Cohort - Ravulizumab to Ravulizumab (N=36) | Extension Period: LN Cohort - Placebo to Placebo (N=18) | Extension Period: IgAN Cohort - Ravulizumab to Ravulizumab (N=42) | Extension Period: IgAN Cohort - Placebo to Ravulizumab (N=23)
COVID-19 (Infections and infestations) | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0
Cardiac failure acute (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Subcutaneous abscess (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Gastroenteritis norovirus (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Tendon rupture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Testis cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Seizure (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Depression (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lupus nephritis (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Epstein-Barr virus infection reactivation (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Soft tissue infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hepatic enzyme increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypertensive crisis (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Nephrotic syndrome (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Initial Evaluation Period: LN Cohort - Ravulizumab (N=38) | Initial Evaluation Period: LN Cohort - Placebo (N=19) | Initial Evaluation Period: IgAN Cohort - Ravulizumab (N=43) | Initial Evaluation Period: IgAN Cohort - Placebo (N=23) | Extension Period: LN Cohort - Ravulizumab to Ravulizumab (N=36) | Extension Period: LN Cohort - Placebo to Placebo (N=18) | Extension Period: IgAN Cohort - Ravulizumab to Ravulizumab (N=42) | Extension Period: IgAN Cohort - Placebo to Ravulizumab (N=23)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Normocytic anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pericarditis (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cushingoid (Endocrine disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Conjunctival haemorrhage (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Optic nerve disorder (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ulcerative keratitis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vitreous floaters (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 6 (9) | 2 (3) | 4 (5) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 6 (6) | 2 (2) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 5 (5) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Mouth ulceration (Gastrointestinal disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Salivary gland enlargement (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 3 (3) | 3 (3) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 4 (4) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza like illness (General disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Malaise (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Peripheral swelling (General disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oedema (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vaccination site pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypertransaminasaemia (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Seasonal allergy (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 4 (4) | 0 (0) | 5 (6) | 1 (1) | 3 (3) | 1 (1) | 6 (6) | 0 (0)
COVID-19 (Infections and infestations) | 3 (3) | 1 (1) | 4 (4) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 3 (4) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 3 (3) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Oral candidiasis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oral herpes (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bacterial infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Conjunctivitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fungal foot infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Localised infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Periodontitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vulvovaginal candidiasis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Immunisation reaction (Injury, poisoning and procedural complications) | 0 (0) | 2 (4) | 0 (0) | 0 (0) | 0 (0) | 1 (4) | 0 (0) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 2 (2) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Activated partial thromboplastin time prolonged (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood magnesium decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Liver function test increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Impaired fasting glucose (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 (3) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 5 (5) | 2 (2) | 0 (0) | 0 (0) | 3 (4) | 1 (1) | 3 (3) | 0 (0)
Sciatica (Nervous system disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tremor (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Nephrotic syndrome (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Menstruation irregular (Reproductive system and breast disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cervical dysplasia (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemorrhagic ovarian cyst (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Postmenopausal haemorrhage (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 6 (7) | 2 (2) | 3 (4) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sputum increased (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 5 (5) | 1 (1) | 0 (0) | 3 (7) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diffuse alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Butterfly rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chronic cutaneous lupus erythematosus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Raynaud's phenomenon (Vascular disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Essential hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
The LN cohort of the study was terminated early due to lack of efficacy.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
There IS an agreement between the Principal Investigator and the Sponsor (or its agents) that restricts the PI's rights to discuss or publish trial results after the trial is completed.

DOCUMENTS (2):
  • Study Protocol (2024-03-26): https://cdn.clinicaltrials.gov/large-docs/39/NCT04564339/Prot_000.pdf
  • Statistical Analysis Plan (2025-04-21): https://cdn.clinicaltrials.gov/large-docs/39/NCT04564339/SAP_001.pdf